CLINICAL TRIAL: NCT03556852
Title: CARBETOCIN VERSUS RECTAL MISOPROSTOL FOR MANAGEMENT OF THIRD STAGE OF LABOR IN WOMEN AT LOW RISK OF POSTPARTUM HEMORRHAGE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed M Maged, MD, professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 38
Record Dates: First submitted 2018-06-04; First posted 2018-06-14 (Actual); Last update posted 2019-10-11 (Actual); Status verified 2019-10

CONDITIONS: Postpartum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — carbetocin; Misoprostol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CARBETOCIN (Active Comparator): received 1 ampoule of Carbetocin (100 μg/ml) added to 10 cc saline and given IV after the delivery of the baby.
  Interventions: Drug: Carbetocin
- MISOPROSTOL (Active Comparator): received 4 rectal misoprostol tablets (800 μg) after the delivery of the baby.
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Carbetocin — 1 ampoule of Carbetocin (100 μg/ml) added to 10 cc saline and given IV after the delivery of the baby
  Arms: CARBETOCIN
Drug: Misoprostol — 2 rectal misoprostol tablets (800 μg) after the delivery of the baby.
  Arms: MISOPROSTOL

SUMMARY:
150 pregnant women admitted for spontaneous, induced or augmented vaginal delivery and categorized as low risk for postpartum hemorrhage (PPH) were divided randomly into two groups. Carbetocin group (C) received 1 ampoule of Carbetocin (100 μg/ml) (Pabal®, Draxis/Multipharma, Egypt, under license from DRAXIS PHARMA-Canada) added to 10 cc saline and given IV after the delivery of the baby. Misoprostol group (M) received 2 rectal misoprostol tablets (800 μg) (Misotac; SIGMA Pharm, Cairo, Egypt) after the delivery of the baby. Blood samples were tested to measure hemoglobin levels upon admission to the labor room and 12 hours after delivery

DETAILED DESCRIPTION:
150 pregnant women admitted for spontaneous, induced or augmented vaginal delivery and categorized as low risk for postpartum hemorrhage (PPH) were divided randomly into two groups. Carbetocin group (C) received 1 ampoule of Carbetocin (100 μg/ml) (Pabal®, Draxis/Multipharma, Egypt, under license from DRAXIS PHARMA-Canada) added to 10 cc saline and given IV after the delivery of the baby. Misoprostol group (M) received 2 rectal misoprostol tablets (800 μg) (Misotac; SIGMA Pharm, Cairo, Egypt) after the delivery of the baby. Blood samples were tested to measure hemoglobin levels upon admission to the labor room and 12 hours after delivery

ELIGIBILITY:
Inclusion Criteria:

singleton pregnancy 36-40 weeks of gestation vertex presentation. normotensive hemoglobinlevel > 10 gm/dl

• Noncomplicated pregnancy

Exclusion Criteria:

* Women with history of Postpartum hemorrhage in previous deliveries uterine fibroids previous cesarean section medical disorders (e.g. diabetes, anemia, coagulation disorders, cardiac, hepatic and renal diseases) antepartum hemorrhage

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 150 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2019-05-24 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
prevention of post partum hemorrhage after vaginal delivery | 24 hours after delivery
  Number of participants experienced postpartum hemorrhage

SECONDARY OUTCOMES:
drugs side effects | 24 hours after delivery
  Number of subjects experienced Hemodynamic changes (blood pressure , pulse and respiratory rate ) , GIT side effects as nausea , vomiting and metallic taste, Vasomotor effects as flushing, headache , itching

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, Principal Investigator — professor
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Maged AM, Waly M, Fahmy RM, Dieb AS, Essam A, Salah NM, Hussein EA, Nabil H. Carbetocin versus rectal misoprostol for management of third stage of labor among women with low risk of postpartum hemorrhage. Int J Gynaecol Obstet. 2020 Feb;148(2):238-242. doi: 10.1002/ijgo.13056. Epub 2019 Dec 2. PMID 31736069